CLINICAL TRIAL: NCT07058935
Title: The Asia-Pacific Mitral & Tricuspid Valve-in-Valve/Valve-in-Ring Registry (AP ViV Registry)
Status: Recruiting | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-4264
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Valve Disease, Heart
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mitral Valve-in-Valve: Patients who have undergone or will undergo a transcatheter mitral valve-in-valve procedure.
- Mitral Valve-in-Ring: Patients who have undergone or will undergo a transcatheter mitral valve-in-ring procedure.
- Tricuspid Valve-in-Valve: Patients who have undergone or will undergo a transcatheter tricuspid valve-in-valve procedure.
- Tricuspid Valve-in-Ring: Patients who have undergone or will undergo a transcatheter tricuspid valve-in-ring procedure.

SUMMARY:
A retrospective and prospective, observational, multicenter cohort study of consecutive patients undergoing transcatheter mitral/tricuspid ViV or ViR procedure with balloon expandable valve across participating sites in Asia-Pacific.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21
2. Had at least one documented Mitral valve-in-valve/valve-in-ring procedure done during the period of 1 Jan 2023 to current date. (Retrospective) OR Planned to undergo a Mitral valve-in-valve/valve-in-ring procedure. (Prospective) OR Had at least one documented Tricuspid valve-in-valve/valve-in-ring procedure done during the period of 1 Jan 2023 to current date. (Retrospective) OR Planned to undergo a Tricuspid valve-in-valve/valve-in-ring procedure. (Prospective)

Exclusion Criteria:

1. Active endocarditis
2. Any other conditions which investigator deems unsuitable for participation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing transcatheter mitral/tricuspid ViV or ViR procedure with balloon expandable valve across participating sites in Asia-Pacific from 1 Jan 2023 to 31 Dec 2035.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | From date of procedure to 10 years

CONTACTS AND LOCATIONS:
Locations (8):
- John Hunter Hospital, New Lambton Heights, Australia
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
- India (2):
  - MGM Healthcare Pvt Ltd, Chennai, Tamil Nadu
  - The Madras Medical Mission, Chennai, Tamil Nadu
- Waikato Hospital, Hamilton, New Zealand
- National Heart Centre Singapore, Singapore, Singapore
- Ramathibodi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No